CLINICAL TRIAL: NCT04810923
Title: Application of Injectable Platelet-Rich Fibrin for the Treatment of Temporomandibular Joint Osteoarthritis: A Randomized Controlled Clinical Trial
Brief Title: Application of Injectable Platelet-Rich Fibrin for the Treatment of Temporomandibular Joint Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-11/47
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; injectable platelet-rich fibrin; Arthrocentesis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthrocentesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-PRF group (Experimental): arthrocentesis procedure plus four consecutive intra-articular injection of i-PRF.
  Interventions: Procedure: i-PRF
- Control group (Experimental): arthrocentesis procedure alone.
  Interventions: Procedure: Arthrocentesis

INTERVENTIONS:
Procedure: i-PRF — intra-articular i-PRF injection after arthrocentesis
  Arms: i-PRF group
Procedure: Arthrocentesis — Arthrocentesis procedure with 2 to 3 mL saline solution to lavage the superior compartment of temporomandibular joint.
  Arms: Control group

SUMMARY:
The authors designed a randomized, controlled, double-blind clinical trial after the ethical approval by the University Ethics Committee. The patients with temporomandibular joint osteoarthritis (TMJ-OA) randomly assigned one of the two treatment groups: intra-articular injection of injectable platelet-rich fibrin (i-PRF) after arthrocentesis procedure as i-PRF group and arthrocentesis procedure alone as control group. The primary outcome variable was pain levels at preoperatively, and postoperatively at 1st, 2nd, 3rd, 6th and 12th month. The secondary outcome variables included maximum mouth opening (MMO), lateral and protrusive movements.

DETAILED DESCRIPTION:
The authors designed a randomized, controlled, double-blind clinical trial after the ethical approval by the University Ethics Committee. The patients with TMJ-OA randomly assigned one of the two treatment groups: intra-articular injection of i-PRF after arthrocentesis procedure as i-PRF group and arthrocentesis procedure alone as control group. All treatment procedures were completed by the same experienced surgeon under the local anesthesia. The procedure of arthrocentesis was performed using the standard technique and after arthrocentesis procedure, the i-PRF injection was performed in the test group.

The primary outcome variable was pain levels at preoperatively, and postoperatively at 1st, 2nd, 3rd, 6th and 12th month. The secondary outcome variables included maximum mouth opening (MMO), lateral and protrusive movements.

ELIGIBILITY:
Inclusion Criteria:

* patients with osteoarthritis (OA) of one or two temporomandibular joint (TMJ)
* maximum mouth opening less than 35 mm
* impeded protrusive and lateral movements
* localized pain of the affected joint

Exclusion Criteria:

* systemic or malignant diseases affecting TMJ-OA assessment
* previous invasive or surgical treatments of TMJ unrelated to OA
* edentulous patients
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Change of Pain Level | at preoperatively, and postoperatively at 1st, 2nd, 3rd, 6th and 12th month
  Pain level was measured with a visual analog scale (VAS) before treatment, and at postoperative follow-up (1st, 2nd, 3rd, 6th and 12th month).

SECONDARY OUTCOMES:
Change of maximum mouth opening | at preoperatively, and postoperatively at 1st, 2nd, 3rd, 6th and 12th month
  Maximum mouth opening was assessed by measuring the distance between the incisal border of upper and lower central incisors
Change of lateral movement | at preoperatively, and postoperatively at 1st, 2nd, 3rd, 6th and 12th month
  Lateral movement was measured from the labioincisal contact between upper central incisors to the same point of lower central incisors
Change of protrusive movement | at preoperatively, and postoperatively at 1st, 2nd, 3rd, 6th and 12th month
  Protrusive movement was measured from the incisal border of upper central incisors to same point of lower central incisors

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Işık, Principal Investigator — Ege University
Locations (1):
- Ege University, Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No